CLINICAL TRIAL: NCT06016179
Title: Phase I Intra-patient Dose Escalation Study of the IL-6 Receptor Antagonist Tocilizumab Delivered Via Pleural and Peritoneal Catheters in Patients With Pleural Effusion or Peritoneal Ascites Due to Metastatic Cancer
Brief Title: Tocilizumab Delivered Via Pleural and Peritoneal Catheters in Patients With Advanced Metastatic Cancer
Acronym: RIOT2
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Allegheny Singer Research Institute (also known as Allegheny Health Network Research Institute) (Other)
Responsible Party: Principal Investigator, Patrick Wagner, MD, FACS, Investigator, Allegheny Singer Research Institute (also known as Allegheny Health Network Research Institute)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023-137
Record Dates: First submitted 2023-07-28; First posted 2023-08-29 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Malignant Pleural Effusion; Malignant Ascites
Keywords: Malignant Pleural Effusion; Malignant Ascites; Tocilizumab; IL-6 receptor antagonist; peritoneal cavity; pleural cavity; intraperitoneal; intrapleural
MeSH Terms: conditions — Pleural Effusion, Malignant | interventions — tocilizumab

STUDY DESIGN:
Intervention Model Description: Intra-patient dose escalation administration of tocilizumab via pleural and peritoneal catheters
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment Arm - intracavitary tocilizumab (Experimental): Four incremental weekly intra-cavitary doses of tocilizumab starting at 0.5μg/mL and increasing to 1.6μg/mL, 5μg/mL and 50μg/mL once a week over four weeks.
  Interventions: Drug: Tocilizumab

INTERVENTIONS:
Drug: Tocilizumab — Each patient will receive four incremental weekly intra-cavitary doses of tocilizumab starting at 0.5μg/mL and increasing to 1.6μg/mL, 5μg/mL and 50μg/mL once a week over four weeks.
  Other Names: Actemra

SUMMARY:
The purpose of this study to find out if tocilizumab can be safely infused into chest or abdominal cavities of patients with malignancy ascites (MA) or malignant pleural effusions (MPE). Patients will have a total of 4 doses, one dose administered each week. Each dose will be greater than the previous one.

DETAILED DESCRIPTION:
This is an open label, Phase 1, intra-patient dose escalation study to determine the feasibility of catheter-based intra-pleural and intra-peritoneal administration of tocilizumab at doses up to 50μg/mL in patients with malignant pleural effusions (MPE) and malignant ascites (MA) and to determine the frequency and type of adverse events.

This study is open to patients who have had or are having chest or abdomen drains placed during cancer treatment to relieve pressure due to buildup of cancerous fluid. Some patients have drains that are temporary (single-use), while others have drains that are left in place (indwelling) for repeated or continuous at-home drainage.

Research participants, in addition to the standard treatment above, will undergo a series of four weekly infusions of the study drug into the body cavities, using the drains to inject the drug. The dose of the drug will be increased at each of the four visits. Each treatment session will last about one hour, and participants donate 12 milliliters (1 tablespoon) of blood before and after the treatment.

Fluid drained from the body cavity, which is normally discarded, will instead be collected for analysis. Researchers will analyze the blood and fluid for markers of your immune system's reaction to the drug. The total study duration is expected to be no more than 10 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females ages 18-89 years
2. Female patients must have a negative pregnancy test and agree to use contraception. Female patients receiving tocilizumab should maintain adequate contraceptive measures during and for a minimum of 90 days after the last dose of tocilizumab. Male patients receiving tocilizumab should maintain adequate contraceptive measures during and for a minimum of 60 days after the last dose of tocilizumab.
3. Biopsy-proven diagnosis of malignancy with cytologic or radiographic evidence of malignant pleural effusion or ascites
4. Scheduled to undergo standard-of-care pleural or peritoneal drainage catheter placement
5. ECOG 0-2
6. Able to read and understand consent in English and provide informed consent

Exclusion Criteria:

1. Pediatric patients
2. Laboratory abnormalities that indicate clinically significant inflammatory process AST/SGOT > 2 times the upper limit of normal ALT/SGPT > 2 times the upper limit of normal Total bilirubin > 2 times the upper limit of normal Creatinine > 2.5 mg/dL Hemoglobin < 7 mg/dL White blood cell count < 3,000/ mm3 Platelet count < 70,000/mm3 Absolute neutrophil cell count < 2,000 per mm3
3. ECOG > 3
4. Subjects who are unable to comply with study procedures including travel for weekly outpatient clinic visits
5. Pregnant and lactating women
6. Active immunotherapy within 30 days; concurrent chemotherapy or targeted therapy is permitted but for patients with a history of prior immunotherapy, the most recent dose should be >30 days prior to the first treatment visit
7. Investigational drug use within 30 days prior to first treatment dose
8. History of systemic autoimmune disease (CRS, GCA, PJIA, RA, and SJIA)
9. Patient with known hypersensitivity to tocilizumab (IL-6)
10. Active infection
11. Medical contraindication or history of adverse reaction to acetaminophen or diphenhydramine

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2024-01-30 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Successful intra-cavitary administration of tocilizumab | 6 weeks
  Number of patients with successful administration of tocilizumab
Adverse Events | 6 weeks
  To identify the frequency and type of adverse events (AE) following intrapleural or intraperitoneal administration of tocilizumab at doses up to 2.5 mg (intrapleural) or 25 mg (intraperitoneal) using CTCAE v5.0

SECONDARY OUTCOMES:
Pharmacokinetics Analysis | 4 weeks
  Measuring serum receptor occupancy levels
Pharmacokinetics Analysis | 4 weeks
  Measuring intracavity fluid receptor occupancy levels
Biomarkers | 4 weeks
  Change in Pleural cytokine concentrations
Biomarkers | 4 weeks
  Change in Peritoneal Cytokine concentrations
Biomarkers | 4 weeks
  Change in immune cell density

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Wagner, MD, Principal Investigator — Director of Complex General Surgical Oncology
Locations (1):
- Allegheny Health Network Cancer Institute, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No